CLINICAL TRIAL: NCT01981109
Title: A Study to Evaluate Characteristics Predictive of a Positive Imaging Study for Distant Metastases in Patients With Castration-Resistant Prostate Cancer
Brief Title: Positive Imaging Study for Distant Metastases in Patients With Castration-Resistant Prostate Cancer
Acronym: PREDICT
Status: Terminated | Type: Observational
Why Stopped: Administrative reasons
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Other Study IDs: P12-1
Record Dates: First submitted 2013-10-28; First posted 2013-11-11 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Castration-Resistant Prostate Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of this research is to describe patient characteristics predictive of an imaging study positive for distant metastases in patients with castration-resistant prostate cancer and no known distant metastases.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to the initiation of study procedures.
* Men ≥ 18 years of age.
* Histologically documented prostatic adenocarcinoma.
* History of Castration-Resistant Prostate Cancer.

Exclusion Criteria:

* Known M1 disease.
* Undergone imaging study for metastatic prostate cancer ≤ 3 months.
* ECOG performance status ≥ 3.
* Known malignant pleural effusions or ascites.
* Current or prior treatment with investigational therapy for M0 Castration-Resistant Prostate Cancer (Taxotere (docetaxel), Provenge® (sipuleucel-T), Zytiga (abiraterone acetate), Xtandi (enzalutamide), Jevtana (cabazitaxel), or Xofigo (radium Ra 223 dichloride).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with Castration-Resistant Prostate Cancerand no known M1 disease who are at least 18 years of age at the time of screening are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Brown, MD, Study Director — Dendreon Pharmaceuticals, LLC
Locations (58):
- United States (58):
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - Urological Associate of Southern Arizona, Tucson, Arizona
  - Sequoia Urology Center, Atherton, California
  - Prostate Oncology Specialist, Inc., Marina del Rey, California
  - Sutter Medical Group, Sacramento, California
  - Genesis Research, San Diego, California
  - Urology Associates of San Luis Obispo, Templeton, California
  - The Urology Center of Colorado, Denver, Colorado
  - Advanced Urology, P.C, Parker, Colorado
  - Howard University Hospital, Washington D.C., District of Columbia
  - Urology Center of South Florida, Miami, Florida
  - Idaho Urologic Institute, Meridian, Idaho
  - Comprehensive Urologic Care, SC, Lake Barrington, Illinois
  - Uro Partners/ RMD Clinical Research, Melrose Park, Illinois
  - Associated Urological Specialists, LLC, Palos Heights, Illinois
  - 1st Urology, PSC, Jeffersonville, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Kansas City Urology Care, PA, Overland Park, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Jewish Hospital, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Mid Atlantic Urology Associates, Greenbelt, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Michigan Institute of Urology, Troy, Michigan
  - Metro Urology, Plymouth, Minnesota
  - Metro Urology, Woodbury, Minnesota
  - Saint Louis VAMS, St Louis, Missouri
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Urology Center Research Institute, Englewood, New Jersey
  - Delaware Valley Urology, LLC, Mount Laurel, New Jersey
  - National Translational Research Group, East Setauket, New York
  - Integrated Medical Professionals, PLLC, North Hills, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Associated Medical Professionals of NY, PLLC, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Durham Veterans Affairs Medical Center, Durham, North Carolina
  - Carolina Urology Partners, Gastonia, North Carolina
  - Central Ohio Urology Group, Gahanna, Ohio
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - Stepherson Cancer Center, Oklahoma City, Oklahoma
  - Portland Veterans Administration Medical Center, Portland, Oregon
  - Oregon Urology Institute, Springfield, Oregon
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Urology Health Specialists, LLC, Bryn Mawr, Pennsylvania
  - Lancaster Urology, Lancaster, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - The Conrad Pearson Clinic, Germantown, Tennessee
  - Tennessee Urology Asociates, Knoxville, Tennessee
  - Urology Associates, P.C., Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - Houston Metro Urology, Houston, Texas
  - UT Memorial Hermann Cancer Center, Houston, Texas
  - Oncology San Antonio Research LLC, San Antonio, Texas
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
  - Medical Oncology Associates, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Sipuleucel-T: A Study to Evaluate Characteristics Predictive of a Positive Imaging Study for Distant Metastases in Patients with Castration-Resistant Prostate Cancer
Period: Overall Study
Arm/Group | Sipuleucel-T
Started | 225
Completed | 1
Not Completed | 224
Not completed — Death | 36
Not completed — Withdrawal by Subject | 40
Not completed — Lost to Follow-up | 9
Not completed — No Discontinuation Documentation | 37
Not completed — Study Termination | 100
Not completed — No data available | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 205
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Total | 77.2 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 225
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Total: American Indian or Alaska Native | 0
  Total: Asian | 0
  Total: Native Hawaiian or Other Pacific Islander | 1
  Total: Black or African American | 51
  Total: White | 173
  Total: More than one race | 0
  Total: Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: Centemeters] | 175.3 (8.3)
Weight [Mean (Standard Deviation); unit: Kg] | 92.7 (20.1)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.2 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Occurrence Measured in Time of an Image Showing Positive for M1 (Metastatic Disease) at Baseline to Registration
Description: The primary endpoint for the study will be the occurrence of an imaging study at baseline that is positive for M1 (yes or no) among all patients in the primary analysis population.The primary analysis population consists of patients who had a current diagnosis of having non metastatic (M0) disease at baseline. These patients underwent imaging scans at baseline and were assessed for metastatic (M1) versus non metastatic (M0) disease.
Time Frame: Each enrolled subject will be evaluated at baseline for the occurrence of metastatic disease by positive imaging scan.
Population: There were 206 patients at baseline that had a valuable data that were assessed. The results were 151 patients that had non-metastatic (M0) and 55 patients that had metastatic disease (M1) disease. The study terminated early therefore no further statistical analysis was performed.
Measure: Mean (Standard Deviation); unit: years
Groups:
- M0- No Distant Metastases; M1-Distant Metastases: A Study to Evaluate Characteristics Predictive of a Positive Imaging Study for Distant Metastases in Patients with Castration-Resistant Prostate Cancer
Arm/Group | M0- No Distant Metastases | M1-Distant Metastases
Number analyzed (Participants) | 151 | 55
years | 10.9 (6.4) | 8.8 (5.9)

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were not collected in this trial as investigational treatment was not administered in this study. Patients received commercial Provenge® (sipuleucel-T), therefore all SAEs were reported to the Safety Reporting group following full prescribing directions.
Description: Adverse Events and Serious Adverse Events were not collected in this trial as investigational treatment was not administered in this study. Patients received commercial Provenge® (sipuleucel-T), therefore all SAEs were reported to the Safety Reporting group following full prescribing directions.
Arm/Group | Sipuleucel-T
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was designed to analyze 1200 patients. Early termination resulted in only 206 patients reporting a definitive diagnosis per imaging scan. Given this much smaller number of patients, the analyses do not provide reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study will be published and/or presented in an integrated manner reflecting the results observed across all participating centers. Accordingly, decisions on timing and content of publications and presentations relating to the Study will be coordinated by Dendreon in communication with institutions contributing patients to the Study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT01981109/Prot_SAP_000.pdf